CLINICAL TRIAL: NCT01246154
Title: An Evaluation of Exercise Tolerance in Asthmatic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Physio Care (Industry)
Responsible Party: MUTHUKUMAR, PHYSIO CARE
Other Study IDs: PC001
Record Dates: First submitted 2010-11-19; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: To Evaluate
Keywords: ASTHMA
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EXERCISE TOLERANCE
  Interventions: Other: EXERCISE TRAINING

INTERVENTIONS:
Other: EXERCISE TRAINING — EXERCISE TRAINING

SUMMARY:
To evaluate exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

- 40-50 YEARS

Exclusion Criteria:

* NO EXCERBATIONS

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: KNOWN ASTHMATIC PATIENTS
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Physio Care, Thanjavur, Tamil Nadu, India